CLINICAL TRIAL: NCT02297984
Title: Changes of Serum Neuroglobin and HIF-1α Concentrations in Early-phase of Acute Ischemic Stroke
Brief Title: Serum Neuroglobin and HIF-1α in Acute Ischemic Stroke
Status: Completed | Type: Observational
Sponsor: Shanghai 6th People's Hospital (Other)
Responsible Party: Principal Investigator, Hao Chen, Doctor, Shanghai 6th People's Hospital
Other Study IDs: H1583-660145
Record Dates: First submitted 2014-11-19; First posted 2014-11-21 (Estimated); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Acute Ischemic Stroke
Keywords: Neuroglobin; HIF-α; Acute ischemic stroke; Prognosis
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute ischemic stroke: Patients who suffered from acute ischemic stroke within 12 hours for the first time before entry into the study.

SUMMARY:
Neuroglobin has shown rich neuroprotective effects against cerebral ischemia and hypoxia, and therefore has the potential to impact outcomes after acute ischemic stroke. Hypoxia inducible factor (HIF)-1α is neuroprotective in several models of experimental brain injury and is increased in brain after acute cerebral infarction in humans and experimental animals.The investigators sought to examine the changes in serum neuroglobin and HIF-1α concentrations in patients with acute ischemic stroke during the initial 96-h period after stroke and assessed the relation between them and the relation of them to prognosis of such patients with acute ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acute ischemic stroke
* Admission within 12 hours

Exclusion Criteria:

* Lacunar infarction
* Cerebral hemorrhagic infarction
* Epilepsy or epileptic persons
* History of neurological diseases, myocardial infarction, renal and hepatic abnormalities and metabolic diseases
* Contraindications to antiplatelet treatments
* Serial blood samples could not be obtained

Ages: 42 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient group comprised 24 male and 16 female. Their age ranged from 42 to 76 years. Locations of infarct, as evidenced by radiologic and neurologic symptoms or signs, included the territories of the middle cerebral artery (13 cases), the posterior cerebral artery (9 cases) the anterior cerebral artery (8 cases), vertebrobasilar area (7 cases), and watershed area (3 cases with cortical and subcortical low densities crossing typical vascular territories).
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2013-10; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Modified Rankin Scale scores | 3 months
  0 = No symptoms; 1 = No significant disability. Able to carry out all usual activities, despite some symptoms; 2 = Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities; 3 = Moderate disability. Requires some help, but able to walk unassisted; 4 = Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted; 5 = Severe disability. Requires constant nursing care and attention, bedridden, incontinent; 6 = Dead.

SECONDARY OUTCOMES:
Glasgow Outcome Scale scores | 3 months
  Glasgow Outcome Scale 1 = death; Glasgow Outcome Scale 2 = vegetative state; Glasgow Outcome Scale 3 = severe neurological deficit; Glasgow Outcome Scale 4 = mild neurological deficit and Glasgow Outcome Scale 5 = premorbid level of functioning or completely recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Lixia Xue, M.D., Ph.D., Study Director — Shanghai 6th People's Hospital
Locations (1):
- Shanghai Sixth People's Hospital, Shanghai, China